CLINICAL TRIAL: NCT06346834
Title: A Study to Evaluate the Immunogenicity and Safety of Sequential Vaccination Among Infants With Poliomyelitis Vaccine (Vero Cells), Inactivated, Sabin Strains （Hereinafter as "sIPV") From Different Manufacturers.
Brief Title: Sequential Vaccination of Poliomyelitis Vaccine (Vero Cells), Inactivated, Sabin Strains From Different Manufacturers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-sIPV-4002
Record Dates: First submitted 2024-01-29; First posted 2024-04-04 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): sIPV: Sinovac Biotech Co., Ltd., Beijing
  Interventions: Biological: sIPV
- control group (Active Comparator): sIPV: Beijing Institute of Biological Products Co., LTD.
  Interventions: Biological: sIPV

INTERVENTIONS:
Biological: sIPV — One dose of the experimental/control vaccine will be administered to 4-month-old infants who have already received two doses of sIPV from Beijing Institute of Biological Products Co., LTD.

SUMMARY:
To evaluate the immunogenicity and safety of sequential vaccination with Sinovac sIPV among infants who have received two doses of Biological Products Co., Ltd. sIPV.

DETAILED DESCRIPTION:
In this study, two hundred infants ≤ 12 months of age vaccinated with two doses of sIPV produced by Beijing Institute of Biological Products Co., Ltd., will be enrolled with a balanced male-to-female ratio. After enrollment with informed consent from the guardians of the participants, they will be divided into two groups, i.e., the study group and the control group, according to the 1:1 ratio. They will be vaccinated with one dose of the sIPV produced by Sinovac or the sIPV produced by Beijing Institute, respectively. The 30-minute observation will be conducted after the vaccination. Immediate reactions will be observed and solicited adverse events within 0-7 days, while unsolicited adverse events within 0-30 days will be collected to evaluate vaccine safety. About 2.5-3.0 ml of venous blood will be collected from all participants before and 30 days after vaccination, and anti-poliovirus type 1, type 2, and type 3 neutralizing antibody tests will be performed to evaluate immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* (1) Healthy infants of ≤ 12 months of age;
* (2) Can provide proof of legal identity;
* (3) Have completed two doses of sIPV vaccination at Beijing Institute;
* (4) Able to provide proof of sIPV vaccination;
* (5) The participant's guardian can understand and agree to sign the informed consent form.

Exclusion Criteria:

* (1) Known severe allergy to vaccines or vaccine components, such as urticaria, dyspnea, angioneurotic edema;
* (2) Received immunoglobulins or other blood products, or plan to receive such treatment during the study;
* (3) Received ≥14 days of immunosuppressive or other immunomodulatory therapy or cytotoxic therapy, or plan to receive such therapy during the study;
* (4) Received another investigational vaccine within 28 days before receiving the study vaccine;
* (5) Received a live attenuated vaccine within 14 days before receiving the trial vaccine;
* (6) Received a subunit or inactivated vaccine within 7 days before receiving the trial vaccine;
* (7) Acute exacerbation of various acute illnesses or chronic diseases within the last 7 days;
* (8) Those who had a fever with an axillary temperature >37.0°C before receiving the study vaccine;
* (9) Participants who, in the judgment of the investigator, have any other factors that make them unsuitable for participation in the study.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Increase (GMI) | 30 days
  -The neutralizing antibody GMI against different types (Type I, II and III) at day 30 after vaccination;
Geometric Mean Titer (GMT) | 30 days
  -The neutralizing antibody GMT against different types (Type I, II and III) at day 30 after vaccination;
Seropositivity rate | 30 days
  -The seropositivity rate of neutralizing antibody against different types (Type I, II and III) at day 30 after vaccination;
Seroconversion rate | 30 days
  -The seroconversion rate of neutralizing antibody against different types (Type I, II and III) at day 30 after vaccination;
Adverse reaction incidence | 30 days
  -The incidence of adverse reaction within 30 days after vaccination;
Serious adverse events incidence | 30 days
  -The incidence of serious adverse events within 30 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Disease Control and Prevention Center, Xiaonan District, Xiaogan City, Xiaogan, China

IPD SHARING:
Plan to Share IPD: No